CLINICAL TRIAL: NCT01379521
Title: A Phase II Randomized, Double-blinded, Multicenter Asian Study Investigating the Combination of Transcatheter Arterial Chemoembolization (TACE) and Oral Everolimus (RAD001, Afinitor®) in Localised Unresectable Hepatocellular Carcinoma (HCC) - The TRACER Study
Brief Title: Safety and Efficacy of RAD001 + TACE in Localized Unresectable HCC
Acronym: TRACER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to low enrollment. This resulted in the study being underpowered and inconclusive.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001OHK02
Record Dates: First submitted 2011-06-01; First posted 2011-06-23 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Localised; unresectable; chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- everolimus + TACE (Experimental): everolimus 7.5mg/day by mouth + transcatheter arterial chemoembolization (TACE)
  Interventions: Drug: everolimus
- placebo + TACE (Placebo Comparator): Placebo by mouth + transcatheter arterial chemoembolization (TACE)
  Interventions: Drug: everolimus placebo

INTERVENTIONS:
Drug: everolimus
  Other Names: RAD001; Afinitor®)
  Arms: everolimus + TACE
Drug: everolimus placebo
  Arms: placebo + TACE

SUMMARY:
This study will evaluate the role of everolimus in combination with local Transcatheter Arterial Chemoembolization (TACE) procedure in patients with localized unresectable Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed hepatocellular carcinoma limited to liver and not suitable for resection, liver transplant, or radiofrequency ablation.
* Intermediate stage (stage B) (according to recognized guidelines) and suitable for TACE therapy
* At least one nodule between > 2cm and ≤ 15cm in diameter with no vascular invasion or abdominal lymph node or distant metastases.
* Must have 1 tumor which can be measured in 1 dimension according to specified criteria (RECIST and mRECIST) and has not previously been treated with any type of therapy.
* ECOG performance status < 2cm
* Cirrhotic status of Child-Pugh class A or early B
* HBV-DNA or HBsAg positive at screen or baseline: preventative treatment with anti-viral started 1-2 weeks prior to receiving study drug

Exclusion Criteria:

* Any local and/or investigational drugs within 28 days prior to randomization
* Active bleeding during the last 28 days prior to screening including variceal bleeding
* Prior therapy with mTOR inhibitors
* Tumor burden of > 60% liver involvement
* Prior systemic or local therapy including TACE except for the first TACE at Day 0), surgery or liver transplantation
* Failed first TACE at Day 0, Cycle 1 for any reason
* Known history of human immunodeficiency virus (HIV) seropositivity (HIV testing is not mandatory)
* Alcohol intake of 80 grams per day
* Undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from surgery
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Novartis Investigative Site, Hong Kong, Hong Kong
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung, Taiwan
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Linkou District
- Novartis Investigative Site, Chiang Mai, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 65 patients who were screened they reflect the actual enrolment but 59 patients were randomized and were included in the FAS, the Safety Set and the PP Set. There were no exclusions. Post-Treatment evaluations included any patients that was treated and does not reflect the number completed in the Overall Study.
Period: Overall Study -Treatment Period
Arm/Group | Everolimus + TACE | Placebo + TACE
Started | 33 | 26
Completed | 0 | 0
Not Completed | 33 | 26
Not completed — Adverse Event | 3 | 0
Not completed — Abnormal test procedure results | 0 | 1
Not completed — Disease Progression | 23 | 22
Not completed — New Cancer Therapy | 1 | 0
Not completed — Protocol Deviation | 0 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Administrative Problems | 1 | 0
Not completed — Death | 2 | 1
Period: Post-Treatment Evaluations
Arm/Group | Everolimus + TACE | Placebo + TACE
Started | 25 | 21
Completed | 0 | 0
Not Completed | 25 | 21
Not completed — Disease Progression | 22 | 20
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + TACE | Placebo + TACE | Total
Number analyzed (Participants) | 33 | 26 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.29) | 61.0 (10.32) | 59.6 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 29 | 19 | 48

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) Based on the Modified RECIST Criteria
Description: Time to Progression (TTP) defined as the time from the date of randomization to the date of first documented radiological confirmation of disease progression based on modified RECIST criteria. Progressive Disease: >20% increase in sum of the longest diameters (SLD) of "viable" target lesion (arterial phase enhancement)
Time Frame: 3, 6, 12, 18 and 24 months
Population: Full Analysis Set (FAS) comprises all randomized patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 33 | 26
months | 6.3 [4.3 to 6.6] | 6.4 [4.0 to 8.9]

2. Secondary Outcome: Overall Response Rate (ORR) and Disease Control Rate (DCR) Based on the Modified RECIST
Description: Overall response rate was defined as the number of patients whose best overall response was either complete response or partial response according to the modified RECIST. Complete response: Disappearance of arterial phase enhance-ment in all target lesions. Partial response: >30% decrease in sum of the longest diameters (SLD) of "viable" target lesion (arterial phase enhance-ment)Disease control rate was defined as the number of patients with a best overall response of complete response, partial response or stable disease. The study was terminated early due to slow enrollment of 4 years, higher than anticipated screen failure rate due to a higher than anticipated proportion of patients having advanced liver disease and a change in clinical practice the total of 80 patients was not reached with only 59 patients recruited in total. The study was underpowered due to termination therefore data was not collected and the outcome measure was not analyzed.
Time Frame: 6, 12 months, end of study
Population: Full Analysis Set (FAS) comprises all randomized patients. The trial results are inconclusive as the study was underpowered due to termination therefore data was not collected and the outcome measure was not analyzed.
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Progression Based on Original RECIST
Description: Time to Progression (TTP) defined as the time from the date of randomization to the date of first documented radiological confirmation of disease progression based on original RECIST criteria. Progressive Disease: >20% increase in sum of the longest diameters (SLD) of target lesions with an absolute increase of ≥5 mm; new lesions. The study was terminated early due to slow enrollment of 4 years, higher than anticipated screen failure rate due to a higher than anticipated proportion of patients having advanced liver disease and a change in clinical practice the total of 80 patients was not reached with only 59 patients recruited in total. The study was underpowered due to termination therefore data was not collected and the outcome measure was not analyzed.
Time Frame: 6, 12 months, end of study
Population: as for outcome 2
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Response Rate (ORR) and Disease Control Rate (DCR) Based on Original RECIST
Description: Overall response rate was defined as the number of patients whose best overall response was either complete response or partial response according to the Complete response: Disappearance of all target lesions or lymph nodes <10 mm in the short axis Partial response: >30% decrease in sum of the longest diameters (SLD) of target lesions Disease control rate was defined as the number of patients with a best overall response of complete response, partial response or stable disease. The study was terminated early due to slow enrollment of 4 years, higher than anticipated screen failure rate due to a higher than anticipated proportion of patients having advanced liver disease and a change in clinical practice the total of 80 patients was not reached with only 59 patients recruited in total. The study was underpowered due to termination therefore data was not collected and the outcome measure was not analyzed.
Time Frame: 6, 12 months, end of study
Population: as for outcome 2
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause. If death had not occurred at the date of the analysis cut-off then OS was censored at the date of the last contact.
Time Frame: 6, 12, 18, 24, 30 months
Population: Full Analysis Set (FAS) comprises all randomized patients. The trial results are inconclusive as the study was underpowered
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 33 | 26
months | 29.9 [12.0 to NA] — The trial results are inconclusive as study was underpowered therefore upper limit was not calculated due to not enough events. | 21.7 [19.4 to 27.9]

6. Secondary Outcome: Incidences of Cumulative New Nodular Recurrence, Portal Vein Invasion and Extra Hepatic Metastases
Description: Incidences of cumulative new nodular recurrence, portal vein invasion and extra hepatic metastases but incidence of portal vein invasion meant those patients without documented vascular invasion at screening/baseline. The study was terminated early due to slow enrollment of 4 years, higher than anticipated screen failure rate due to a higher than anticipated proportion of patients having advanced liver disease and a change in clinical practice the total of 80 patients was not reached with only 59 patients recruited in total. The study was underpowered due to termination therefore data was not collected and the outcome measure was not analyzed.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With a Decrease in the Sum of the of Longest Diameters (SLD) of Target Lesions From Baseline to 30 Months
Description: Percentage of participants with a decrease in the sum of the of longest diameters (SLD) of target lesions from Baseline to 30 months
Time Frame: baseline, 30 months
Population: Full Analysis Set (FAS) comprises all randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus + TACE | Placebo + TACE
Number analyzed (Participants) | 32 | 25
Percentage of participants | 93.8 | 88.0

ADVERSE EVENTS:
Arm/Group | Everolimus + TACE | Placebo + TACE
Serious Adverse Events (participants affected / at risk) | 10/33 | 7/26
Other Adverse Events (participants affected / at risk) | 33/33 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + TACE (N=33) | Placebo + TACE (N=26)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Liver abscess (Infections and infestations) | 1 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Post embolisation syndrome (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + TACE (N=33) | Placebo + TACE (N=26)
Anaemia (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 19 | 17
Abdominal pain upper (Gastrointestinal disorders) | 8 | 5
Ascites (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Gastritis (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 9 | 2
Nausea (Gastrointestinal disorders) | 6 | 5
Stomatitis (Gastrointestinal disorders) | 7 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6
Mucosal inflammation (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 5 | 0
Pyrexia (General disorders) | 12 | 12
Hepatitis b (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 7 | 5
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Hypertension (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.